CLINICAL TRIAL: NCT05057377
Title: Estimating Highest Capacity Performance During Evaluation of Walking for Individuals With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0300
Record Dates: First submitted 2021-08-18; First posted 2021-09-27 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-TBI Participants: Over a 2-day period post-TBI adults age 18 years and older, will undergo overground assessments with a questionnaire regarding motivation during day 1, followed by robotic safety-environment assessments during day 2.
  Interventions: Diagnostic Test: Standard Overground Assessment; Diagnostic Test: Robotic Safety-Environment Assessment

INTERVENTIONS:
Diagnostic Test: Standard Overground Assessment — The standard overground methods to assess three main components of walking are the 10 Meter Walk Test (meters/second, used to measure speed), 5x Sit-to-Stand (seconds, used to measure strength), and the 6-Minute Walk Test (meters, used to measure endurance).
Diagnostic Test: Robotic Safety-Environment Assessment — The methods for assessment of the three main components of walking in the robotic environment will be the maximum walking speed tolerated (meters/second, to measure speed), deadband resistance (kilograms, to measure strength), and the 6-minute walk test (meters, to measure endurance).

SUMMARY:
Traumatic brain injury (TBI) due to trauma and/or neurologic disease is a leading cause of long-term disability in the United States. The loss of balance for people with a traumatic brain injury can have a large effect on their walking abilities and this can come with a number of challenges. There is a greater risk of falling after being discharged from the hospital. In addition, people are more likely to become sedentary after TBI, which leads to the loss of muscle strength.

To help provide the best care, clinicians need accurate measurements when people begin their therapy, as well as throughout to ensure they are making appropriate progress. The tests currently used by clinicians may not provide the most accurate measurements that show what a person is capable of physically doing. The study you are being asked to participate in aims to provide more accurate measurements by using a robotic treadmill device and by assessing motivating factors that are important to you. The treadmill device will allow us to more accurately test your walking ability in a safe, fall-free environment.

DETAILED DESCRIPTION:
Traumatic brain injury due to trauma and/or neurologic disease is a leading cause of long-term disability in the United States. Balance impairments observed within the post-TBI population can greatly impact walking abilities and pose a variety of challenges. Following hospital discharge, there is a greater fall risk as well as a decrease in physical activity and increase in sedentary behaviors that lead to deconditioning.

It is difficult to determine the extent of what a person is capable of doing using current overground assessment methods, which are the current standard means of physical capability measurements (i.e. 6-minute walk test, 5 times sit-to-stand, 10-meter walk test). Improvement of walking and balance outcomes in this population requires the re-evaluation of current approaches and the testing/implementation of new approaches. This will allow more appropriate assessment of baseline walking abilities in order to apply the appropriate amount of challenge during rehabilitation training. This study will involve the use of a robotic treadmill device in order to determine maximum walking capacities of participants and compare these capacities to standard overground assessments. It has been shown that walking speeds overground are correlated with walking speeds on a robotic device (and even specifically on the KineAssist-MX, which will be used for this project). If it is found that maximum capacities be greater on the robotic device, rehabilitation training goals can be more appropriately tailored to these participants.

The aims and hypotheses of this research project are:

Aim 1) Assess function at preferred performance in an overground environment vs. a safety-enhanced robotic environment to establish concurrent validity.

Hypothesis 1) Participants with the highest overground performances (strength, speed, and endurance) will have the highest performances on the KineAssist-MX and vice versa.

Aim 2) Assess maximum capacities of participants over ground vs. in the safety-enhanced robotic environment to establish content validity.

Hypothesis 2) Maximum capacity will be higher in the safety-enhanced robotic environment than overground and vice versa. Therefore, people will be able to do more in the robotic environment than overground.

Aim 3) Assess the capacities of individuals across different baseline functional strata to establish usability.

Hypothesis 3) Individuals in the lower quadrants of baseline function will have lower maximum capacities in the safety-enhanced robotic environment.

This study will occur over a two-day period of time during which participants will undergo overground assessments during day 1 and robotic safety-environment assessments during day 2. There will be no interventions implemented.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 years and older
* All demographic groups will be invited to participate and would have equal access
* Post-TBI individuals currently enrolled at the Moody Neurorehabilitation Institute
* Ambulatory with or without assistive devices
* Subjects with expressive aphasia in the case of a caregiver able to provide assistance when needed
* English-speaking only
* Medically stable (controlled hypertension, no arrhythmia, stable cardiovascular status)
* Able to provide written informed consent

Exclusion Criteria:

* Subjects with loss of lower limb
* History of serious cardiac disease (e.g., myocardial infarction)
* Uncontrolled blood pressure (systolic pressure >140 mmHg, diastolic blood pressure >90 mmHg)
* Subjects with receptive aphasia
* Presence of cerebellar and brainstem deficits
* Severe cognitive disorder
* Uncontrolled respiratory or metabolic disorders
* Major or acute musculoskeletal problems
* Spasticity management that included phenol block injections within 12 months or botulinum toxin injections within 4 months of the study
* Participants undergoing any rehabilitation therapy during the timeframe of this study.
* Body weight greater than 250 pounds (due to robotic device weight restrictions)
* Non-English speaking individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, post-TBI individuals currently enrolled at the Moody Neurorehabilitation Institute.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in 10-Meter Walk Test-Overground | Baseline, pre-intervention.
  The 10-meter walk test assess walking speed in meters per second over a short duration.
Change in 5x Sitting to Standing Resistance Test | Baseline, pre-intervention.
  In order to measure walking strength, participants will be asked to perform a Sit-to-Stand test. Beginning from a sitting position, a participant is asked to stand and return to a seated position. They will be asked to repeat this procedure 5 times.
6-Minute Walk Test | Baseline, pre-intervention.
  In order to measure walking endurance, participants will be asked to walk as far as they are able to comfortably walk during a 6 minute time period, with the total distance (in meters) being the outcome.
Top Walking Speed/Max Tolerated using Robotic Device | During the intervention.
  In order to measure walking speed, and with the assistance of the safety enhanced robotic-treadmill device, a participant's maximum walking speed will be measured in meters per second.
Deadband Resistance/Max Tolerated using Robotic Device | During the intervention.
  In order to measure walking strength, participants will be asked to walk on the robotic-treadmill device as fast as they can over a series of trials. Resistance of the treadmill will be increased until a maximum is reached and recorded.
6-Minute Walk Test using Robotic Device | During the intervention.
  In order to measure walking endurance, participants will be asked to walk as far as they are able to comfortably walk during a 6 minute time period while using the robotic-treadmill device.

CONTACTS AND LOCATIONS:
Overall Officials: David Brown, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- Moody Neurorehabilitation Institute at Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided